CLINICAL TRIAL: NCT04143672
Title: A Cohort Study on Association Between Pain Sensitivity by Pain Sensitivity Questionnaire and Postoperative Opioid Requirement
Brief Title: Pain Sensitivity Questionnaire and Postoperative Opioid Requirement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SNUH-HJ-1
Record Dates: First submitted 2019-10-27; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; pain sensitivity
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): The following tests will be performed on the study subjects.
  1. Pain catastrophizing scale
  2. Hospital Anxiety and Depression scale-Anxiety Subscale (HADS-A)
  3. Pain sensitivity questionnaire
  4. Pain pressure threshold using electronic digital pressure algometer
  Interventions: Device: Electronic digital pressure algometer; Diagnostic Test: Pain sensitivity questionnaire

INTERVENTIONS:
Device: Electronic digital pressure algometer — Evaluation of pain threshold using an algometer is conducted one day before surgery.
  The pressure of the plunger of algometer is applied vertically to the patient's right thenar muscle belly at a speed of 10 N/sec by the tester. Then the tester removes the algometer when the patients start to feel pain and record the pressure recorded on the algometer.
  Other Names: electronic digital pressure algometer (FGN-20B, Shimpo, Kyoto, Japan)
Diagnostic Test: Pain sensitivity questionnaire — Evaluation of pain threshold using the Korean-version pain sensitivity questionnaire is conducted one day before surgery.

SUMMARY:
This study aims to investigate the potential association between pain sensitivity questionnaire score, the severity of postoperative pain, and postoperative analgesic requirement in patients with open colorectal cancer surgery. This information may be used to guide the optimal postoperative pain management, and ultimately improve patient's quality of life.

DETAILED DESCRIPTION:
We plan to investigate the predictive ability of the PSQ as well as experimental parameters of pain sensitivity using electronic algometer and other known risk factors for postoperative pain in 100 patients scheduled for open colorectal cancer surgery.

The following items are investigated before surgery; Age, sex, level of education, type of surgery, past surgical history, presence of chronic pain, the expected maximal pain score (VAS) after surgery, Pain catastrophizing scale, anxiety scale (HADS-A), Pain sensitivity questionnaire, and pain threshold measured by electronic algometer.

The total opioid consumption is investigated for 24 and 48 hours after surgery. In addition, the severity of postoperative pain is measured by the 11-point VAS at 24 and 48 hours after surgery. Patient satisfaction with postoperative pain control is also investigated at 48 hours after surgery using the 7-point patient's satisfaction scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Patients scheduled for open colorectal cancer surgery under general anesthesia
* ASA status I-III
* Ability to read and understand the information sheet, questionnaires, and the - consent form
* Patients scheduled for using IV-PCA after surgery

Exclusion Criteria:

* Unable to read and understand the information sheet, questionnaires, and the consent form
* Severe medical or psychological diseases
* Patients with preoperative chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Total fentanyl consumption during 24 hours | postoperative 24 hours
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia
Total fentanyl consumption during 48 hours | postoperative 48 hours
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia

SECONDARY OUTCOMES:
Postoperative pain score | postoperative 24, 48 hours
  11-pointed NRS pain score at resting/coughing/movement NRS (0-10): 0, "no pain"; 10, "worst pain imaginable"
Patient satisfaction for postoperative pain management | postoperative 48 hours
  7-pointed likert scale (very satisfied-somewhat satisfied-satisfied-neutral-dissatisfied-somewhat dissatisfied-very dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jintae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital